CLINICAL TRIAL: NCT04996186
Title: Symptoms and Treatment Assessment of Ano-Rectal Disorders in Multiple Sclerosis Patients : STAR-Q (STAR Questionnaire): Validation of a New Tool to Better Explore and Manage Bowel Dysfunction.
Brief Title: Symptoms and Treatment Assessment of Ano-Rectal Disorders in Multiple Sclerosis Patients : STAR-Q
Acronym: STAR-Q
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Clinical Professor, Head of neurourology department, APHP, Tenon Hospital, Paris, France, Pierre and Marie Curie University
Other Study IDs: GRC 01 GREEN STAR Q
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis; Constipation; Fecal Incontinence
Keywords: multiple sclerosis; constipation; fecal incontinence; questionnaire; evaluation; quality of life
MeSH Terms: conditions — Multiple Sclerosis; Constipation; Fecal Incontinence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patients with Multiple sclerosis, with an age older than 18 years old and symptoms of fecal incontinence or chronic constipation
  Interventions: Other: Clinical interviews

INTERVENTIONS:
Other: Clinical interviews — Semi-qualitative interviews and questionnaire STAR-Q
  Other Names: Semi-qualitative interviews and questionnaire

SUMMARY:
Multiple sclerosis (MS) is known to cause urinary disorders, sexual and bowel dysfunction. Urinary symptoms due to MS are well known and profit of multiple questionnaire or tool developed in MS patients.

Prevalence of bowel disorders in MS is difficult to assess. Some studies up to 70% bowel disorders in MS patients. Constipation and fecal incontinence are the two main symptoms in neurogenic bowel dysfunction and frequently coexist in this population, generally in association with urinary disorders.

Because of the high prevalence of bowel disorders their and the major impact on the quality of life of patients with Multiple sclerosis (PwMS) , and the cross-talk bladder-rectum (persistence of anorectal dysfunction leading to poor neurogenic bladder control) assessment of bowel disorders in MS is necessary. But this evaluation is difficult as no specific score exist. The neurogenic Bowel Dysfunction score (NBD) is often used. The NBD was developed and validated for spinal cord injury (SCI) population but not for PwMS MS. Yet NBD is often used in research for all neurologic patients despite its lack of sensibility in various neurogenic population other than spinal cord injury patient. As recommended in a Cochrane revue in 2014, there is a need of a specific evaluation for bowel symptoms in neurogenic population, especially for PwMS.

The aim of the study was to create and validate a new multidimensional questionnaire to assess bowel dysfunction and impact on quality of life in patients with MS.

The investigators conducted a prospective multicenter study (8 centers) between June 2019 to April 2021. This study was developed in 3 steps. First step was literature review and qualitative interview. Then the second step was the feasibility study to evaluate comprehension, acceptability of the different items. The last part of the study was the validation study of the questionnaire. This part of the study was performed between June2020 and April 2021. Validation study allowed to determine the psychometric properties of the new tool.

Patients aged over 18 years with multiple sclerosis diagnosed on the 2017 revised McDonald's criteria were included. Patients not able to read or understand the objectives and procedures for conducting the protocol and patient who had a recent relapse of MS were excluded.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune autoimmune central nervous system (CNS) disorder characterized by demyelinisation and central neurologic damage. MS is the first cause of disability in young adults and affects 2.8 million people in the world.

Multiple sclerosis (MS) is known to cause urinary disorders, sexual and bowel dysfunction. Urinary symptoms due to MS are well known and profit of multiple questionnaire or tool developed in MS patients.

Prevalence of bowel disorders in MS is difficult to assess. Some studies up to 70% bowel disorders in MS patients. Constipation and fecal incontinence are the two main symptoms in neurogenic bowel dysfunction and frequently coexist in this population, generally in association with urinary disorders. Chronic constipation and fecal incontinence were defined by Rome IV criteria. According to these criteria, constipation is a bowel disorder in which symptoms of difficult, infrequent, or incomplete defecation predominate for at least 3 months and fecal incontinence is defined as the recurrent uncontrolled passage of fecal material for at least 3 months.

Moreover, neurogenic bowel dysfunction has a real impact on quality of life and can cause social isolation.

Because of the high prevalence of bowel disorders their and the major impact on the quality of life of patients with Multiple sclerosis (PwMS) , and the cross-talk bladder-rectum (persistence of anorectal dysfunction leading to poor neurogenic bladder control) assessment of bowel disorders in MS is necessary. But this evaluation is difficult as no specific score exist. The neurogenic Bowel Dysfunction score (NBD) is often used. The NBD was developed and validated for spinal cord injury (SCI) population but not for PwMS MS. Yet NBD is often used in research for all neurologic patients despite its lack of sensibility in various neurogenic population other than spinal cord injury patient. As recommended in a Cochrane revue in 2014, there is a need of a specific evaluation for bowel symptoms in neurogenic population, especially for PwMS.

The aim of the study was to create and validate a new multidimensional questionnaire to assess bowel dysfunction and impact on quality of life in patients with MS.

The investigators conducted a prospective multicenter study (8 centers) between June 2019 to April 2021. This study was developed in 3 steps. First step was literature review and qualitative interview. Then the second step was the feasibility study to evaluate comprehension, acceptability of the different items. The last part of the study was the validation study of the questionnaire. All these phases allowed a full psychometric validation of the questionnaire.

Patients aged over 18 years with multiple sclerosis diagnosed on the 2017 revised McDonald's criteria were included. Patients not able to read or understand the objectives and procedures for conducting the protocol and patient who had a recent relapse of MS were excluded.

Step 1: literature review and qualitative interview. The investigators conducted a review of literature on Pubmed to know all the existing questionnaires or tools developed and validated to assess neurogenic bowel dysfunction in MS. All articles published until April 2020 were included. The following keywords were used: "neurogenic bowel dysfunction", "constipation", "fecal incontinence", "anorectal disorders", "multiple sclerosis".

In addition a single trained nurse performed qualitative interviews with patients suffering from ano rectal disorders secondary to MS. These interviews were lead in two phases. First part allowed to determine the wording of the different symptoms and mode of response for each item. The second part of the face-to-face was free and patients could express themselves if there was a gap in our list of symptoms.

During this first phase of the study a panel of 8 experts was selected, composed of neuro urologists and gastro enterologists.

The first version of the questionnaire was made based on the patients' qualitative interviews, on the reactions and comments of the expert team and on the literature review.

Step 2: Feasibility study The feasibility study was conducted between April 2020 and June 2020. This pilot study included 30 patients and was performed to assess comprehension, acceptability and pertinence of the items the investigators have created to build the questionnaire. More of response was also evaluate by patients.

Step 3: Validation study. This part of the study was performed between June2020 and April 2021. Validation study allowed to determine the psychometric properties of the new tool. All items were discussed for ceil or floor effect by the expert team. Each item with more than 50% of patients having the same response were discussed by panel experts to decide if they were excluded or not of the final version.

To obtain good psychometric properties, the investigators included 10 patients for each items of the questionnaire in the final version. This number of subjects was calculated to allow univariate and multivariate logistic regression.

Internal consistency reliability was calculated using the alpha coefficient of Cronbach. Each response has been transformed in a numeric value to perform this test. Alpha coefficient of Cronbach was considered as very good if > 0.7.

Test-retest reliability was tested using the intraclass correlation coefficient (ICC) which was significant over 0.7. The first questionnaire was filled at the end of the first consultation and patients had to mail a second questionnaire (filled at home) 7 to 14 days after the first consultation.

Statistical analyses: Final version of STAR-Q (Symptoms and Treatment Assessment of Ano-Rectal disorders in multiple sclerosis patients Questionnaire) was composed by 3 sub domains. First one was symptoms, second one was treatment, and a third sub domain was quality of life.

For each sub domains, the investigators calculated an alpha coefficient of Cronbach and a ICC. the investigators also assessed these properties for total score.

Total score was compared to NBD total score which represents gold standard in ano rectal disorders and thus constitutes the reference testing external consistency. Finally, PGI (Patient Global Improvment) severity scores were used to determine category of severity for STAR-Q scores.

All statistical analyzes were performed with the R-studio version 3.3.1 and Statviews (SAS institute V 5.0).

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple sclerosis diagnosed on the 2017 revised McDonald's criteria
* over 18 years old

Exclusion Criteria:

* inability to read and to understand the questions
* recent relapse of multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting or hospitalized in a rehabilitation center or in a neuro-urology center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Reproductibility of STAR-Q | 1 day
  Patients were asked to answer a second time the questionnaire with a second evaluation at 14 days after the first one. The "intra-class correlation coefficient" (ICC) was used to determine if these evaluations could lead to similar results for each question. An ICC > 0.70 was necessary to define reproducibility.
Acceptability and comprehension of STAR-Q | 1 day
  Each patient was asked to rate each version of the 22 questions with a four-point Likert scale (A: perfect, B: good, C: average, D: bad) regarding acceptance and comprehension of the questions.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PHD, Principal Investigator — Sorbonne Université, GRC 001, GREEN, AP-HP, Hôpital Tenon, F-75020, Paris, France
Locations (1):
- Department of Neuro- Urology, Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided